CLINICAL TRIAL: NCT01625338
Title: An Open-Label Study of GS-7977 + Ribavirin With or Without Peginterferon Alfa-2a in Subjects With Chronic HCV Infection Who Participated in Prior Gilead HCV Studies
Brief Title: Open-Label Study of Sofusbuvir+Ribavirin With or Without Peginterferon Alfa-2a in Subjects With Chronic HCV Infection Who Participated in Prior Gilead HCV Studies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-334-0109; 2012-000571-16 (EudraCT Number)
Record Dates: First submitted 2012-06-07; First posted 2012-06-21 (Estimated); Results first posted 2015-11-09 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Hepatitis C
Keywords: HCV genotype 2 (GT-2); HCV genotype 3 (GT-3); HCV; Sustained Virologic Response; Direct Acting Antiviral; Combination Therapy; GS-7977; Ribavirin; Open Label
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SOF+RBV 12 Weeks (Experimental): SOF+RBV for 12 weeks
  Interventions: Drug: SOF; Drug: RBV
- SOF+RBV 24 Weeks (Experimental): SOF+RBV for 24 weeks
  Interventions: Drug: SOF; Drug: RBV
- SOF+RBV+Peg-IFN 12 Weeks (Experimental): SOF+RBV+Peg-IFN for 12 weeks
  Interventions: Drug: SOF; Drug: RBV; Drug: Peg-IFN

INTERVENTIONS:
Drug: SOF — SOF 400 mg tablet administered orally once daily
  Other Names: Sovaldi®; GS-7977; PSI-7977
Drug: RBV — RBV tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
Drug: Peg-IFN — Peg-IFN 180 μg administered once weekly by subcutaneous injection
  Arms: SOF+RBV+Peg-IFN 12 Weeks

SUMMARY:
This study will evaluate the efficacy, safety, and tolerability of sofosbuvir (SOF; GS-7977) in combination with ribavirin (RBV) with or without pegylated interferon (Peg-IFN) in adults with chronic hepatitis C virus (HCV) infection who participated in a prior Gilead HCV study and have not achieved sustained virologic response (SVR).

ELIGIBILITY:
Inclusion Criteria:

* Infection with HCV
* Must have participated in a prior Gilead HCV study
* Use of highly effective contraception methods if female of childbearing potential or sexually active male
* Eligible patients include those in the following

  * received placebo or Peg-IFN+RBV in a control arm
  * previously participated in a Gilead-sponsored HCV study and did not attain sustained virologic response 24 weeks after discontinuation of therapy (SVR24) on a regimen containing:

    * Sofosbuvir+RBV
    * Peg-IFN and/or RBV in combination with one or more Gilead investigational direct-acting agents

Exclusion Criteria:

* Pregnant or nursing female or male with pregnant female partner
* Current or prior history of clinical hepatic decompensation
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
* Chronic use of systemically administered immunosuppressive agents
* Active drug abuse
* Use of any prohibited concomitant medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2012-06; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bittoo Kanwar, MD, Study Director — Gilead Sciences
Locations (174):
- United States (67):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Franco Felizarta, MD, Bakersfield, California
  - Arrowhead Regional Medical Center, Colton, California
  - Southern California Transplantation Institute, Research Foundation Liver Center, Coronado, California
  - eStudy Site, La Mesa, California
  - Kaiser Permanente, Los Angeles, California
  - Lightsource Medical/Peter J. Ruane MD, Inc., Los Angeles, California
  - California Liver Institute, Los Angeles, California
  - Anthony Mills MD, Inc., Los Angeles, California
  - eStudySite, Oceanside, California
  - University of California Davis Medical Center, Sacramento, California
  - University of California, San Diego, California
  - Resarch and Education, Inc., San Diego, California
  - Medical Associates Research Group, San Diego, California
  - Kaiser Permanente, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - University of Colorado Hospital, Aurora, Colorado
  - South Denver Gastroenterology, PC, Englewood, Colorado
  - Whitman-Walker Health, Washington D.C., District of Columbia
  - Pointe West Infectious Diseases d/b/a Bach and Godofsky Infectious Diseases, Bradenton, Florida
  - University of Florida, Gainesville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - University of Miami Center for Liver Diseases, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - Advanced Research Institute, Trinity, Florida
  - South Florida Center of Gastroenterology, PA., Wellington, Florida
  - Atlanta Gastroenterology Associates, LLC, Atlanta, Georgia
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Gastointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - Digestive Disease Associates, PA, Baltimore, Maryland
  - Johns Hopkins University, Lutherville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Infectious Disease and The Research Institute, Springfield, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Orlando Clinical, Novi, Michigan
  - Minnesota Gastroenterology, P.A., Saint Paul, Minnesota
  - Kansas City Gastroenterology and Hepatology, Kansas City, Missouri
  - ID Care, Inc., Hillsborough, New Jersey
  - AGA Clinical Research Associates, LLC, Township, New Jersey
  - The Gastroenterology Group of South Jersey, Vineland, New Jersey
  - Binghamton Gastroenterology Associates, PC, Binghamton, New York
  - North Shore University Hospital, Manhasset, New York
  - Weill Cornell Medical College, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Clinical Study Center of Asheville, LLC, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Carolinas Center for Liver Disease, Statesville, North Carolina
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Gastro One, Germantown, Tennessee
  - Memphis Gastroenterology Group, PC, Germantown, Tennessee
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Annette C. and Harold C. Simmons Transplant Center, Dallas, Texas
  - Research Specialists of Texas, Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Metropolitan Research, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Bon Secours Saint Mary's Hospital of Richmond, Newport News, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
- Australia (15):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Gallipoli Medical Research Foundation, Greenslopes, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Austin Hospital, Heidelberg, Victoria
  - Monash Medical Centre, Melbourne, Victoria
  - B2 Clinic, Fremantle, Western Australia
  - Canberra Hospital, Australian Capital Territory
  - St. Vincent's Hospital, Fitzroy
  - Royal Brisbane & Women's Hospital, Herston
  - St George Hospital, Kogarah
  - Royal Prince Alfred Hospital, Camperdown, NSW
  - Royal Perth Hospital, Perth Western Australia
  - Princess Alexandra Hospital, State of Queensland
  - Box Hill Hospital, Victoria
- Austria (3):
  - Medizinische Universität Graz, Graz
  - Medizinische Universität Wien, Vienna
  - Wilhelminenspital, Vienna
- Canada (11):
  - University of Calgary, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver Infectious Disease Research and Care Centre, Vancouver, British Columbia
  - Gastrointestinal Research Institute (GIRI), Vancouver, British Columbia
  - John Buhler Research Center, Winnipeg, Manitoba
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Toronto Digestive Diseases Associates, Inc, Vaughan, Ontario
  - Hopital St. Luc, Montreal, Quebec
  - Gordon & Leslie Diamond Health Care Centre, Vancouver
- Remedis s.r.o., Nestátní zdravotnické zarízení, Prague, Czechia
- Estonia (2):
  - West Tallinn Central Hospital, Tallinn
  - Tartu University Hospital, Tartu
- France (14):
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - CHU Estaing, Clermont-Ferrand
  - Hôpital Beaujon, Clichy
  - Hôpital Henri Mondor, Créteil
  - Hôpital Claude Huriez- Service d'Hépato-Gastroentérologie, Lille
  - Hôpital Saint Joseph, Marseille
  - Hopital Saint Eloi, Montpellier
  - Service Hepatologie, Nice
  - Hôpital Saint-Antoine, Paris
  - Groupe Hospitalier Pitié-Salpétrière, Paris
  - Hôpital Haut-Lévêque, CHU Bordeaux, Pessac
  - Centre Hospitalier Universitare de Rennes, Hôpital Pontchaillou, Rennes
  - Centre Hospitalier Universitaire de Strasbourg, Strasbourg
  - Hopital de I'Archet 2, Vandœuvre-lès-Nancy
- Germany (16):
  - Leber- und Studienzentrum am Checkpoint, Berlin
  - Campus Virchow Klinikum, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Klinikum und Fachbereich Medizin Johann Wolfgang Goethe-Universität Frankfurt am Main, Frankfurt am Main
  - PraxisZentrum für Gastroenterologie und Endokrinologie, Freiburg im Breisgau
  - Asklepios Klinik Sankt Georg Hamburg, Hamburg
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Medizinische Universitätsklinik IV (Krehl Klinik) Abt. Gastroenterologie und Infektionskrankheiten, Heidelberg
  - Gastroenterologische Gemeinschaftspraxis, Herne
  - Leberstudienzentrum Kiel, Kiel
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum der Universität München, Munich
  - Centrum fur Interdisziplinare Medizin, Münster
  - Universitatsklinikum Wurzburg, Würzburg
- Italy (10):
  - Casa Sollievo della Sofferenza Hospital, San Giovanni Rotonda, Foggia
  - Ospedale S. Annunziata, Florence
  - Ente Ospedaliero Ospedali Galliera di Genova, Genoa
  - Azienda Ospedaliera Ospedale Niguarda Ca' Granda, Milan
  - Fondazione IRCCS CA Granada - Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera de Padova, Padua
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Fondazione PTV - Policlinico Tor Vergata, Roma
  - I.N.M.I L. Spallanzani IRCCS, Rome
  - Azienda Ospedaliero Universitaria S. Giovanni Battista di Torino, Turin
- Netherlands (3):
  - Academisch Medisch Centrum, Amsterdam
  - Radboud University Nijmegen Medical Centre (UMC St Radboud), Nijmegen
  - Academic Hospital Rotterdam Erasmus Medical Center, Rotterdam
- New Zealand (7):
  - Auckland Clinical Studies, Grafton, Auckland
  - Tauranga Hospital, Tauranga, BOP
  - Christchurch Hospital, Christchurch, Christchurch
  - Wellington Hospital, Newtown, WGN
  - Auckland City Hospital, Auckland
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
- Poland (5):
  - Klinika Chorob Zakaznych i Hep, Bialystok
  - Oddzial Kliniczny Chorob Zakaznych, Chorzów
  - WSSzpital im.Dr.Wj.Bieganskieg, Lodz
  - ID Clinic, Mysłowice
  - Sp Zoz Wojewódzki Szpital, Warsaw
- Fundacion De Investigacion De Diego, San Juan, PR, Puerto Rico
- Spain (7):
  - Hospital Casa de la Maternidad, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Carlos III, Madrid
  - Hospital Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Nuestra Señora de Valme, Seville
  - Hospital General Universitario de Valencia, Valencia
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Skånes Universitetssjukhus, Malmö, Malmo
  - Karolinska University Hospital Huddinge, Stockholm
- United Kingdom (9):
  - The Liver Unit, Paddington, London
  - University of Birmingham, Birmingham
  - Southampton University Hospital, Hampshire
  - London Royal Hospital, GHU, London
  - King's College Hospital, London
  - Chelsea and Westminster Hospital NHS Foundation Trust, London
  - Royal Free Hospital and University College London Hospital, London
  - North Manchester General Hospital, Manchester
  - Nottingham University Hospitals-NHS, Nottingham

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 152 study sites from their prior Gilead study in North America, Europe, Australia, and New Zealand. The first participant was screened on 22 June 2012. The last study visit occurred on 22 December 2014.
Pre-assignment Details: 585 participants were screened.
Groups:
- SOF+RBV 12 Weeks: Sofosbuvir (SOF) 400 mg tablet once daily + ribavirin (RBV) tablets (1000 or 1200 mg daily based on weight) for 12 weeks
- SOF+RBV 24 Weeks: SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 24 weeks
- SOF+RBV+Peg-IFN 12 Weeks: SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) + pegylated interferon (Peg-IFN) 180 µg administered subcutaneously once weekly for 12 weeks in participants
Period: Overall Study
Arm/Group | SOF+RBV 12 Weeks | SOF+RBV 24 Weeks | SOF+RBV+Peg-IFN 12 Weeks
Started | 114 | 200 | 220
Completed | 82 | 156 | 181
Not Completed | 32 | 44 | 39
Not completed — Enrolled but not Treated | 0 | 0 | 1
Not completed — Efficacy Failure | 27 | 39 | 31
Not completed — Lost to Follow-up | 3 | 3 | 2
Not completed — Investigator Decision | 0 | 2 | 1
Not completed — Subject Withdrew Consent | 1 | 0 | 2
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Study Discontinued by Sponsor | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were enrolled and received at least 1 dose of study drug.
Groups:
- SOF+RBV 12 Weeks: SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks
- SOF+RBV+Peg-IFN 12 Weeks: SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) + Peg-IFN 180 µg administered subcutaneously once weekly for 12 weeks in participants
- Total: Total of all reporting groups
Arm/Group | SOF+RBV 12 Weeks | SOF+RBV 24 Weeks | SOF+RBV+Peg-IFN 12 Weeks | Total
Number analyzed (Participants) | 114 | 200 | 219 | 533
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (9.6) | 52 (7.6) | 53 (10.0) | 53 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 50 | 60 | 164
  Male | 60 | 150 | 159 | 369
Race/Ethnicity, Customized [Number; unit: participants]
  White | 105 | 184 | 187 | 476
  Black Or African American | 4 | 2 | 20 | 26
  Asian | 2 | 6 | 8 | 16
  Other | 1 | 3 | 2 | 6
  Not Permitted | 0 | 2 | 2 | 4
  American Indian Or Alaska Native | 2 | 1 | 0 | 3
  Native Hawaiian Or Other Pacific Islander | 0 | 2 | 0 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 19 | 12 | 20 | 51
  Not Hispanic or Latino | 95 | 187 | 197 | 479
  Not Permitted | 0 | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 77 | 82 | 121 | 280
  United Kingdom | 3 | 10 | 8 | 21
  Spain | 1 | 8 | 2 | 11
  New Zealand | 4 | 30 | 6 | 40
  Canada | 7 | 13 | 10 | 30
  Austria | 1 | 2 | 1 | 4
  Netherlands | 2 | 4 | 4 | 10
  Sweden | 2 | 5 | 3 | 10
  Czech Republic | 0 | 0 | 1 | 1
  Poland | 0 | 1 | 8 | 9
  Italy | 3 | 7 | 4 | 14
  Australia | 9 | 14 | 19 | 42
  France | 2 | 10 | 11 | 23
  Germany | 2 | 12 | 18 | 32
  Estonia | 1 | 2 | 3 | 6
HCV Genotype [Number; unit: participants]
  Genotype 1 | 0 | 2 | 134 | 136
  Genotype 2 | 62 | 10 | 8 | 80
  Genotype 3 | 52 | 180 | 74 | 306
  Genotype 4 | 0 | 7 | 3 | 10
  Indeterminate | 0 | 1 | 0 | 1
Cirrhosis Status [Number; unit: participants]
  No | 89 | 138 | 183 | 410
  Yes | 25 | 62 | 36 | 123
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 38 | 59 | 47 | 144
    CT | 61 | 103 | 127 | 291
    TT | 13 | 35 | 40 | 88
    Missing | 2 | 3 | 5 | 10
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.3 (0.87) | 6.4 (0.70) | 6.4 (0.64) | 6.4 (0.72)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 30 | 44 | 36 | 110
  ≥ 800,000 IU/mL | 84 | 156 | 183 | 423

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 25 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 12 Weeks | SOF+RBV 24 Weeks | SOF+RBV+Peg-IFN 12 Weeks
Number analyzed (Participants) | 114 | 200 | 219
percentage of participants | 71.9 | 77.5 | 82.6

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 24 weeks
Population: Safety Analysis Set: participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 12 Weeks | SOF+RBV 24 Weeks | SOF+RBV+Peg-IFN 12 Weeks
Number analyzed (Participants) | 114 | 200 | 219
percentage of participants | 0.9 | 1.0 | 3.7

3. Secondary Outcome: Percentage of Participants With SVR at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR 24 were defined as HCV RNA < LLOQ at 4 and 24 weeks after stopping study treatment, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 12 Weeks | SOF+RBV 24 Weeks | SOF+RBV+Peg-IFN 12 Weeks
Number analyzed (Participants) | 114 | 200 | 219
percentage of participants
  SVR4 | 73.7 | 81.5 | 87.2
  SVR24 | 71.9 | 76.0 | 82.6

4. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as
  * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
  * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
  * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
Time Frame: Up to 24 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 12 Weeks | SOF+RBV 24 Weeks | SOF+RBV+Peg-IFN 12 Weeks
Number analyzed (Participants) | 114 | 200 | 219
percentage of participants | 0.9 | 0.5 | 0

5. Secondary Outcome: Percentage of Participants With Viral Relapse
Description: Viral relapse was defined as HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values or last available posttreatment measurement.
Time Frame: Up to Posttreatment Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 12 Weeks | SOF+RBV 24 Weeks | SOF+RBV+Peg-IFN 12 Weeks
Number analyzed (Participants) | 113 | 199 | 219
percentage of participants | 25.7 | 20.6 | 16.4

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | SOF+RBV 12 Weeks | SOF+RBV 24 Weeks | SOF+RBV+Peg-IFN 12 Weeks
Serious Adverse Events (participants affected / at risk) | 4/114 | 11/200 | 4/219
Other Adverse Events (participants affected / at risk) | 92/114 | 167/200 | 194/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV 12 Weeks (N=114) | SOF+RBV 24 Weeks (N=200) | SOF+RBV+Peg-IFN 12 Weeks (N=219)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Meningitis aseptic (Infections and infestations) | 0 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Myelitis transverse (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Affective disorder (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Mania (Psychiatric disorders) | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Social stay hospitalisation (Social circumstances) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV 12 Weeks (N=114) | SOF+RBV 24 Weeks (N=200) | SOF+RBV+Peg-IFN 12 Weeks (N=219)
Anaemia (Blood and lymphatic system disorders) | 13 | 12 | 26
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 11
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 38
Abdominal pain (Gastrointestinal disorders) | 6 | 7 | 5
Diarrhoea (Gastrointestinal disorders) | 7 | 14 | 28
Nausea (Gastrointestinal disorders) | 22 | 27 | 52
Vomiting (Gastrointestinal disorders) | 7 | 7 | 9
Asthenia (General disorders) | 5 | 9 | 19
Chills (General disorders) | 2 | 3 | 19
Fatigue (General disorders) | 33 | 66 | 97
Influenza like illness (General disorders) | 6 | 5 | 45
Pain (General disorders) | 2 | 4 | 17
Pyrexia (General disorders) | 5 | 1 | 27
Nasopharyngitis (Infections and infestations) | 9 | 22 | 4
Upper respiratory tract infection (Infections and infestations) | 7 | 9 | 2
Decreased appetite (Metabolism and nutrition disorders) | 3 | 8 | 32
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 21 | 37
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 11 | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 17 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 9 | 45
Dizziness (Nervous system disorders) | 4 | 13 | 23
Dysgeusia (Nervous system disorders) | 3 | 0 | 12
Headache (Nervous system disorders) | 15 | 57 | 71
Anxiety (Psychiatric disorders) | 6 | 11 | 14
Depression (Psychiatric disorders) | 7 | 21 | 14
Insomnia (Psychiatric disorders) | 18 | 34 | 37
Irritability (Psychiatric disorders) | 5 | 27 | 38
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 11 | 33
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 12 | 11
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 12
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 14 | 17
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 23 | 40
Rash (Skin and subcutaneous tissue disorders) | 13 | 19 | 35

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years